CLINICAL TRIAL: NCT01213719
Title: Effects of Betaine Supplementation Combined or Not With Creatine Supplementation on Muscle Creatine Content and Strength
Brief Title: Effects of Betaine Supplementation on Strength and Muscle Creatine Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: betaine supplementation
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Subjects
Keywords: betaine, creatine, strength
MeSH Terms: interventions — Creatine; Betaine; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- creatine (Experimental): will receive creatine monohydrate (20g/d) throughout 10 days
  Interventions: Dietary Supplement: creatine
- betaine (Experimental): will receive betaine (2g/d) throughout 10 days
  Interventions: Dietary Supplement: betaine
- placebo (dextrose) (Placebo Comparator): will receive dextrose(20g/d)throughout 10 days.
  Interventions: Dietary Supplement: dextrose
- creatine plus betaine (Active Comparator): will receive creatine (20g/d) plus betaine (2g/d) throughout 10 days
  Interventions: Dietary Supplement: creatine plus betaine

INTERVENTIONS:
Dietary Supplement: creatine — 20g/d throughout 10 days
  Arms: creatine
Dietary Supplement: betaine — 2g/d throughout 10 days
  Arms: betaine
Dietary Supplement: dextrose — dextrose (placebo), 20 g/d throughout 10 days
  Arms: placebo (dextrose)
Dietary Supplement: creatine plus betaine — creatine (20g/d) plus betaine (2g/d) throughout 10 days
  Arms: creatine plus betaine

SUMMARY:
It has been suggested that betaine supplementation may improve muscle strength by increasing muscle creatine content. However, there is no data supporting this assumption. The investigators speculate that betaine supplementation could enhance intramuscular creatine content, which would result in strength improvements.

ELIGIBILITY:
Inclusion Criteria:

* physically inactive
* non-obese

Exclusion Criteria:

* skeletal muscle disturbance
* cardiovascular disturbance
* use of dietary supplements

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
strength | after 10 days

SECONDARY OUTCOMES:
intramuscular creatine content | after 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, PhD, Study Director — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil